CLINICAL TRIAL: NCT00431379
Title: Treatment of Acute Respiratory Distress Syndrome With Tenecteplase: A Dose Escalation Pilot Study: Phase I
Brief Title: Treatment of Acute Respiratory Distress Syndrome With Tenecteplase: A Dose Escalation Pilot Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: drug has expired, no enrollments in study. Company pulled funding
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H0605329
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2013-11

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase

SUMMARY:
The pathogenesis of ARDS appears to be from damage to the alveolar-capillary barrier, which is composed of the microvascular endothelium and the alveolar epithelium. This damage may occur from direct or indirect lung injury. The mechanism of injury to the alveolar capillary barrier appears to be through neutrophil-mediated injury, pro-inflammatory cytokines, ventilator-induced lung injury with alveolar over distention and abnormalities of the coagulation system. This results in blood clot formation in the microcirculation of the lung. Thrombolytics can dissolve blood clots and result in increased blood flow to the organs. This treatment may benefit ARDS patients, thus the purpose of this study.

Hardaway, et al.studied the effects of thrombolytics on ARDS in pigs. The experimental group showed improved oxygenation and survival as compared to controls. There was no bleeding complications noted with this therapy. Dr. Hardaway followed this animal study with a phase I clinical trial involving 20 patients with ARDS. The patients were treated with IV streptokinase or urokinase. Nineteen of the 20 patients showed an increase in PA02 after thrombolytic therapy. There were no significant bleeding complications in patients that were critically ill on ventilators.

We propose an additional phase I pilot study to evaluate the effectiveness and safety of Tenecteplase for the treatment of ARDS. Unlike the other fibrinolytics studied in this disease state, Tenecteplase, is more fibrin specific and has increased resistance to plasminogen activator inhibitor (PAI-I) at greater levels than other available fibrinolytics. We have chosen an experimental dose escalation trial design of tenecteplase that has demonstrated initial safety trends in a Phase I acute ischemic stroke trial. The initial dose is 0.1 mg/kg IV and will increase to 0.2 mg/kg, 0.3 mg/kg, with a final cohort of patients receiving 0.4 mg/kg. Drug administration will be a single dose bolus in each cohort. Advancement of dose will occur if safety is not in question in the previous cohort. We hope this will provide an acceptable benefit risk ratio as the mortality of ARDS is approximately 30 - 60%. All patients will be closely monitored for any change in clotting parameters and signs of bleeding. Tenecteplase will be administered via a peripheral IV as described in the package insert.

DETAILED DESCRIPTION:
1. Treatment of acute respiratory distress syndrome with tenecteplase, a dose escalation pilot study: phase I
2. The study sample size will be 20 patients. The 20 patients will be divided into 4 groups with 5 patients in each group or cohort. The first cohort will received 0.1mg/kg of tenecteplase as a bolus via peripheral IV as described by the package insert and will be closely monitored for safety and efficacy. If there are no adverse events associated with tenecteplase, the second cohort of patients will be enrolled and will receive 0.2 mg/kg of tenecteplase IV bolus. If there are no safety issues, we will proceed with the next cohort at 0.3 mg/kg with a final cohort of patients receiving 0.4 mg/kg of tenecteplase IV bolus. Advancement of dose will occur if safety is not in question in the previous cohort.
3. Tenecteplase will be given as a bolus via peripheral IV as described by package insert.
4. Treatment will be initiated after informed consent is obtained and only >12 hrs after any subcutaneous Heparin has been stopped and >12 hrs after placement of a pulmonary artery catheter, central line or arterial line. Only patients meeting criteria for ARDS (see inclusion criteria) will be considered for the study.
5. Pretreatment assessment: We will obtain informed consent, demographic data, physical examination and medical history, vital signs, PT, PTT, INR, ABG, hemoglobin hematocrit, liver enzymes, cardiac enzymes, creatinine, fibrinogen, fibrin split products, platelets, urine pregnancy test, EKG, chest x-ray, cardiac profile from Swan-Ganz catheter and ventilator settings before treatment begins.
6. Assessment during treatment: Blood samples will be taken every 6 hours for 24 hours and analyzes for PT, PTT, INR, fibrinogen, fibrin split products, platelets, hemoglobin, and hematocrit. Arterial blood gas samples will be taken at hour 1, 2, 3, and every six hours until 24 hours post-injection. Cardiac profile, vital signs and ventilator settings will be monitored at hour 1, 2, 3, and every six hours until 24 hours post-infusion. Adverse events will be monitored every hour for 24 hours.
7. Follow-up assessment: 72 hours post treatment physical exam, vital signs, weight, adverse events, cardiac profile, ventilator settings, PT, PTT, INR, fibrinogen, fibrin split products, platelets, ABG, hemoglobin and hematocrit, liver enzymes, cardiac enzymes, creatinine, EKG and chest x-ray will be obtained. Thirty days post treatment physical exam, vital signs, weight, mortality, adverse events will be followed.
8. Patients will be monitored for signs of clinical bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for full duration of the study by family member.
* Patient-related considerations - See exclusion criteria
* Disease-related considerations - ARDS is indicated by respiratory failure of acute onset, bilateral lung infiltrates, PaO2/Fi02 <200 mmHg,pulmonary artery wedge pressure < 18 mmHg, and need for a ventilator. (If the wedge pressure is >18, the patient is excluded from this study).
* Only acute stage ARDS patients will be enrolled in the study. This is defined by patients with ARDS for <1 week.

Other considerations

* Satisfactory recruitment and cooperation
* A signed informed consent document
* No participation in another clinical and/or observational trial
* No previous participation in this study
* Not a prisoner or otherwise in custody and not institutionalized for mental incompetence.
* Patients with major trauma will only be included 5 days after trauma has occurred.

Exclusion Criteria:

* Bleeding - active internal bleeding
* History of cerebrovascular accident
* Intracranial neoplasm, arteriovenous malformation, or aneurysm or acute trauma
* Known bleeding diathesis
* Severe uncontrolled HTN
* Thrombin time over 2 times laboratory normal
* Prothrombin time or partial thromboplastin time > 2 times normal
* Fibrinogen <100
* Platelets <100
* Creatine >2.0
* Liver function tests > 2 times normal
* History of coagulopathy, ulcer, or stroke
* Systolic blood pressure >180, diastolic blood pressure >110
* History of fibrinolytic use within one month prior to treatment
* History of diabetic retinopathy
* Pregnancy, pregnancy will be ruled out in women of childbearing age by urine test.
* Obstetric delivery or intracranial injury within one month prior to treatment
* Major trauma, major surgery, or CPR within 5 days or minor surgery or minor trauma within 2 days. The classification of major or minor is made by attending physician.
* Patients undergoing non-operative management of liver, spleen, and kidney trauma.
* Aspirin therapy >650mg q day
* Epidural or spinal catheter within 5 days.
* Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, and subacute bacterial endocarditis.
* Over the age of 75 years
* Patients on Xigris

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Survival to Discharge
Safety Analysis of Bleeding Complications

SECONDARY OUTCOMES:
Improved Pa02/Fi02 ratio
Improved cardiac profile
Incidence of organ failure
Decreased ventilator days
Decreased ICU days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis W. Ashley, MD, FACS, Principal Investigator — Medical Center of Central GA; Debra M Kitchens, RN, CEN, Study Chair — Medical Center of Central Georgia
Locations (1):
- Medical Center of Central GA, Macon, Georgia, United States